CLINICAL TRIAL: NCT03624179
Title: Study of Some Risk Factors for Developing Rheumatoid Arthritis
Brief Title: Study of Some Risk Factors for Developing RA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebtesam mostafa, principle investigator, Assiut University
Other Study IDs: AssiutU9
Record Dates: First submitted 2018-07-11; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis patients: complete blood count, Erythrocyte sedimentation rate, C reactive protien ,rheumatoid factor,Anti cyclic citrullinated peptide antibody
- healthy control: complete blood count, Erythrocyte sedimentation rate, C reactive protien ,rheumatoid factor,Anti cyclic citrullinated peptide antibody

SUMMARY:
Introduction Rheumatoid arthritis (RA), a chronic autoimmune disease of unknown etiology, .If not managed early , RA can result in irreversible, painful, and disabling joint damage. RA is often diagnosed using predefined criteria that necessitate clinical, laboratory, and radiologic examinations.

The prevalence of RA among adults is approximately 1-2% affecting women two to four times more often than men.Although RA risk increases with age, it can manifest at any stage of life, including childhood, adolescence, and adulthood.(1-4)( Karlson EW, Mandl LA, Hankinson SE, Grodstein F, Karlson EW, Mandl LA, Hankinson SE, Grodstein F., Karlson EW, Mandl LA, Hankinson SE, Grodstein F, Karlson EW, Mandl LA, Hankinson SE, Grodstein F) To date, a limited number of RA risk or protective factors have been identified, with genetic predisposition to autoimmune response (eg, HLA-DR4 gene) and repeated environmental exposures (eg, tobacco smoke) playing a major role.(3)(Karlson EW, Mandl LA, Hankinson SE, Grodstein F) Heritability of RA is well-established because the lifetime risk of RA and related autoimmune diseases (namely, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, Sjo¨gren's syndrome, and hypothyroidism) increases 1.5 to 3 times in children of women diagnosed with RA.

DETAILED DESCRIPTION:
Patients will answer the following the questationnaire:

Name age gender

1 Socio echonomic status (average salary \year) (Education) (Job) (residence)

1. Body mass index (height\wt2)
2. Disease duration in months.
3. Smoking (yes) (No) Passive smoker Ex smoker
4. Reproductive history:

   * age of menarche….
   * menstrual cycle….. regular or not……. P / C
   * How many pregnancies…….. living.

     * Abortion.
   * patient age at first birth (….).
   * breast feeding…..(yes)…….(no)
   * use of contraceptives (yes)…pills injections IUD (N0)……
   * Does patient get pregnant during disease?...(Yes)……(no)….. Does the arthritis improved (…)or got worse (…..) -flared during the purpurium.(yes) … (No)
   * age of menupause…. 10 Exposure to sun….(yes)…..(No) 11 -Theraputic history… (Newly diagnosed)

     * (Previously diagnosed),
   * Does the patient receiving ttt? (yes) (Steroid)……. (NSAIDS)……. (2nd line drugs) (.Methotrexat(.…), Leflonamide (….) Hydroquine(….) (NO)……..
   * The study will include 100 patients fullfilling ACR 2010
   * Patients well subjected to

     * Through clinical examination with emphysis on joints examination
     * venous blood sampling will withdrawn and the following investigations will be done.
     * Serum VIT D level
     * Serum calcium and phosphorus
     * Anti cyclic citrullinated peptide.
     * ESR

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatoid arthritis diagnosed based on american collegue of rheumatology 2010 criteria with no history of vit D therapy

Exclusion Criteria:

* patients with rheumatoid arthritis on vit D supplements
* patient refusal
* patient not fullfill american collegue of rheumatology 2010 citeria for diagnosis pf rheumatoid arthritis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-20 (Estimated)

PRIMARY OUTCOMES:
vitamin D level | one month
  blood sample using ELISA kits
Body mass index | one month
  weight in kg/m^2

SECONDARY OUTCOMES:
Anti cyclic citrullnated peptide antibodies | one month
  blood sample using ELISA
Rheumatoid factor antibody | one month
  blood sample

REFERENCES:
- [Background] Almodovar PI. Dermatology diagnosis. Tuberculoid leprosy. Bol Asoc Med P R. 1986 Dec;78(12):514-5. No abstract available. PMID 3468952
- [Background] Jankosky C, Deussing E, Gibson RL, Haverkos HW. Viruses and vitamin D in the etiology of type 1 diabetes mellitus and multiple sclerosis. Virus Res. 2012 Feb;163(2):424-30. doi: 10.1016/j.virusres.2011.11.010. Epub 2011 Nov 20. PMID 22119899
- [Background] Ginns LC, Ryu JH, Rogol PR, Sprince NL, Oliver LC, Larsson CJ. Natural killer cell activity in cigarette smokers and asbestos workers. Am Rev Respir Dis. 1985 Jun;131(6):831-4. doi: 10.1164/arrd.1985.131.6.831. PMID 4003932
- [Background] Hodges GR, Loker EF Jr. Letter: Fatal pneumonia cause: avirulent wild-type ADV-7 or vaccine strain ADV-7. Chest. 1975 Jun;67(6):740. No abstract available. PMID 165046
- [Background] Mendes EN, Queiroz DM, Rocha GA, Nogueira AM, Carvalho AC, Lage AP, Barbosa AJ. Histopathological study of porcine gastric mucosa with and without a spiral bacterium ("Gastrospirillum suis"). J Med Microbiol. 1991 Dec;35(6):345-8. doi: 10.1099/00222615-35-6-345. PMID 1753392
- [Result] Karlson EW, Mandl LA, Hankinson SE, Grodstein F. Do breast-feeding and other reproductive factors influence future risk of rheumatoid arthritis? Results from the Nurses' Health Study. Arthritis Rheum. 2004 Nov;50(11):3458-67. doi: 10.1002/art.20621. PMID 15529351
- [Result] Kawakami M, Watanabe N, Ogawa H, Kato A, Sando H, Yamada N, Murase T, Takaku F, Shibata S, Oda T. Cachectin/TNF kills or inhibits the differentiation of 3T3-L1 cells according to developmental stage. J Cell Physiol. 1989 Jan;138(1):1-7. doi: 10.1002/jcp.1041380102. PMID 2783422
- [Result] Merlino LA, Cerhan JR, Criswell LA, Mikuls TR, Saag KG. Estrogen and other female reproductive risk factors are not strongly associated with the development of rheumatoid arthritis in elderly women. Semin Arthritis Rheum. 2003 Oct;33(2):72-82. doi: 10.1016/s0049-0172(03)00084-2. PMID 14625816
- [Result] Cooper GS, Bynum ML, Somers EC. Recent insights in the epidemiology of autoimmune diseases: improved prevalence estimates and understanding of clustering of diseases. J Autoimmun. 2009 Nov-Dec;33(3-4):197-207. doi: 10.1016/j.jaut.2009.09.008. Epub 2009 Oct 9. PMID 19819109
- [Result] Clowse ME, Chakravarty E, Costenbader KH, Chambers C, Michaud K. Effects of infertility, pregnancy loss, and patient concerns on family size of women with rheumatoid arthritis and systemic lupus erythematosus. Arthritis Care Res (Hoboken). 2012 May;64(5):668-74. doi: 10.1002/acr.21593. PMID 22344961
- [Result] Padyukov L, Silva C, Stolt P, Alfredsson L, Klareskog L. A gene-environment interaction between smoking and shared epitope genes in HLA-DR provides a high risk of seropositive rheumatoid arthritis. Arthritis Rheum. 2004 Oct;50(10):3085-92. doi: 10.1002/art.20553. PMID 15476204
- [Result] Reckner Olsson A, Skogh T, Wingren G. Comorbidity and lifestyle, reproductive factors, and environmental exposures associated with rheumatoid arthritis. Ann Rheum Dis. 2001 Oct;60(10):934-9. doi: 10.1136/ard.60.10.934. PMID 11557649